CLINICAL TRIAL: NCT00003029
Title: Infusional 5-Fluorouracil With or Without Cisplatin and With or Without Chronomodulation Against Locally-Advanced or Metastatic Pancreatic Cancer. A Multicenter Randomized Phase III Trial.
Brief Title: Fluorouracil With or Without Cisplatin in Treating Patients With Advanced or Metastatic Cancer of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-05962; EORTC-05962
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Fluorouracil

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells. It is not yet known whether fluorouracil plus cisplatin are more effective than fluorouracil alone in treating patients with metastatic cancer of the pancreas.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil with or without cisplatin in treating patients who have advanced or metastatic cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Confirm the value of chronomodulated infusion with respect to survival in patients with locally advanced or metastatic pancreatic cancer.
* Test the value of adding cisplatin to fluorouracil in extending survival in these patients.

OUTLINE: This is a multicenter, randomized study.

The study design is a 2 X 2 factorial such that patients are allocated to one of 4 treatment groups involving the use or absence of chronomodulation and cisplatin (CDDP). Treatment in each of the 4 groups is repeated for 3 courses where each course is a 5-day course of treatment.

Patients in the first group receive a chronomodulated schedule based on delivery of fluorouracil (FU). Patients in the second group receive a chronomodulated schedule of FU and CDDP. Patients in the third and fourth experimental groups receive flat schedules of FU alone or FU and CDDP, respectively. Dosages of FU are increased across the three courses whereas dosages of CDDP remain constant.

Treatment is continued until disease progression, severe toxicity, or complete remission for more than 4 months occurs.

PROJECTED ACCRUAL: 200 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or cytologic proof of adenocarcinoma of the exocrine pancreas or of a metastasis associated with a radiologically identified pancreatic tumor
* Locally advanced and/or metastatic pancreatic cancer
* No measurable or evaluable target lesion is required
* No brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 40%-100%

Hematopoietic:

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 3 times normal

Renal:

* Creatinine no greater than 1.24 mg/dL OR
* Creatinine clearance at least 80 mL/min

Cardiovascular:

* No overt cardiac disease

Other:

* No peripheral neuropathy
* No uncontrolled infectious or chronic disease
* No second primary except in situ carcinoma of the cervix, or basal or squamous cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunologic therapy

Chemotherapy:

* No prior chemotherapy allowed

Endocrine therapy:

* No concurrent hormonal therapy
* At least 2 weeks since corticoid treatment

Radiotherapy:

* No prior radiotherapy allowed except as an analgesic treatment on metastasis

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 1997-05; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Levi, MD, PhD, Study Chair — Institut de Cancerologie et D'Immunogenetique at Hopital Paul-Brousse
Locations (19):
- Belgium (2):
  - Hopital de Jolimont, Haine-Saint-Paul
  - Les Cliniques Saint-Joseph ASBL, Liège
- France (14):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - Hopital Perpetuel Secours, Levallois-Perret
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Notre-Dame de Bon Secours, Metz
  - Centre Hospitalier de Montlucon, Montluçon
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Saint-Louis, Paris
  - Hopital Cochin, Paris
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Bellevue, Saint-Etienne
  - Clinique de l'Orangerie, Strasbourg
  - Hopital Paul Brousse, Villejuif
- Wolfson Medical Center, Holon, Israel
- Universita G.D'Annunzio Di Chieti, Chieti, Italy
- Hospital Fernando Fonseca, Amadora, Portugal